CLINICAL TRIAL: NCT02857361
Title: An Open Label, Two-way Crossover Study to Evaluate the PK Effects of Two Different Wafer Administration Protocols in Healthy Volunteers Under Fasted Conditions.
Brief Title: Crossover Study to Evaluate the PK Effects of Two Different Wafer Administration Protocols.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: iX Biopharma Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KET011
Record Dates: First submitted 2016-08-02; First posted 2016-08-05 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A: Simultaneous Administration (Experimental): Sublingual ketamine 50mg (2 x 25mg wafers) administered simultaneously at T=0 minute.
  Interventions: Drug: Sublingual ketamine wafers
- Treatment B: Sequential Administration (Experimental): Sublingual ketamine 50mg (2 x 25mg wafers) administered sequentially, one 25 mg wafer at T=0 minute and one 25 mg wafer at T=3 minutes.
  Interventions: Drug: Sublingual ketamine wafers

INTERVENTIONS:
Drug: Sublingual ketamine wafers — Two sublingual ketamine 25 mg wafers
  Other Names: Wafermine

SUMMARY:
The study will look at whether it is preferable to administer two wafers simultaneously or separately.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18-65 years.
* Good general health without clinically significant renal, hepatic, cardiac or respiratory disease, as determined by the Principal Investigator.
* Willing and able to give informed consent and agree to complete all study procedures.
* Have suitable venous access for blood sampling.
* Female participants are eligible only if all the following apply:

  1. Not pregnant (women of child bearing potential must have a negative serum pregnancy test at screening and negative urine pregnancy test at check-in for each inpatient period);
  2. Not lactating;
  3. Not planning to become pregnant during the study;
  4. Be surgically sterile (irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or have undergone bilateral tubal ligation; or be at least two years post-menopausal; or is practicing double-barrier contraception or is using an insertable, injectable, transdermal, or combination oral contraceptive for greater than 2 months prior to screening visits and commits to the use of an acceptable form of highly effective birth control for the duration of the study and for 30 days after the last dose study drug administration.
* BMI within the range of 19-30 kg/m2 (inclusive).
* Deemed able to read and understand English in order to communicate with research staff and complete protocol required questionnaires and forms.

Exclusion Criteria:

* Has a laboratory value at the Screening Visit that is outside the normal range, unless it is judged by the Investigator as not clinically significant after appropriate evaluation. One repeat of initial laboratory testing is allowed.
* AST, ALT and ALP tests in excess of 1.5 times the upper limit of normal.
* Any gastrointestinal condition that could affect drug absorption.
* History of any clinically significant condition involving the bladder or urinary tract, including frequent urinary tract infections (e.g. > 2 per year), or current symptoms of bladder irritation such as frequent or urgent need to urinate or burning with urination.
* History (within the last six months) of or current clinically significant psychiatric disorder including anxiety, psychosis or depression.
* Current inflammatory or ulcerative disease of the oral cavity that could impair the absorption of sublingual medication.
* History of severe allergic or anaphylactic drug-related reactions.
* History of hypersensitivity to ketamine or any of the excipients of Wafermine™.
* Intake of any prescribed or Over-The-Counter (OTC)/non-prescribed drugs, vitamins, supplements or herbal medicines, within 2 weeks of administration of investigational product (or longer if the medication has a half-life long enough to potentially expose the healthy participant to any significant systemic exposure). Exception: Hormone replacement therapy and oral contraceptives in female participants is allowed.
* Use of drugs with enzyme-inducing properties, such as rifampicin and St John's Wort, within 3 weeks or 5 half-lives, whichever is greater, prior to treatment period 1 and throughout the study, or any drug known to be a strong inhibitor of CYP3A4 within 5 half-lives of treatment period 1 and throughout the study.
* Participation in another clinical trial of an investigational agent within 30 days of screening.
* Positive serology for hepatitis C virus (HCV), hepatitis B or human immunodeficiency virus (HIV).
* Clinically significant, as determined by the Investigator, abnormal ECG (12-lead) or vital signs at the screening visit or pre-dose on any treatment day.
* Known or suspected drug (including analgesic drugs or tranquilizers) or alcohol abuse or dependence, as defined by DSM-IV, and not in full remission, as judged by the Investigator, or history of alcohol abuse or excessive intake of alcohol, defined as regular weekly intake of >15 units for men and >10 units for women. (1 unit = 25 mL spirits, 125 mL wine, 250 mL beer or lager.)
* Positive results on the urine drug screen or breath alcohol test at screening and/or pre-dose. A positive result on the urinary drug screen at screening is allowed at the discretion of the Investigator provided the result can be reliably explained by recent medication and/or dietary history.
* Significant history of illicit drug use (as determined by the Investigator).
* Any alcohol use within 24 hours prior to each inpatient treatment period.
* Unwillingness or inability to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the participant returning for subsequent visits on schedule.
* Blood donation (1 unit or more) within 1 month prior to the screening visit and until the end of study participation.
* Current or previous tobacco user (within 12 months prior to screening).
* Participants who routinely consume more than four standard caffeinated beverages per 24-hour period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Bioavailability | 10 hours
  Plasma concentrations collected for 10 hours after simultaneous wafer administration and sequential wafer administration

SECONDARY OUTCOMES:
Number of treatment related adverse events | From time of initial dose until 3 days after final dose.
Participant Acceptance | 20 minutes
  Participant will rate their experience by completing a questionnaire 20 minutes after each dose.
Administrator Acceptance | 20 minutes
  The person administering drug will rate their experience by completing a questionnaire 20 minutes after each dose.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Salman, MD, Principal Investigator — iX Biopharma
Locations (1):
- Linear Clinical Research, Nedlands, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No